CLINICAL TRIAL: NCT01580345
Title: Effect of Docosa-Hexanoic Acid (DHA) Supplements During Pregnancy on Newborn Outcomes in India (DHANI)
Brief Title: Effect of Docosa-Hexanoic Acid (DHA) Supplements During Pregnancy on Newborn Outcomes in India.
Acronym: DHANI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre for Chronic Disease Control, India (Other)
Collaborators: Department of Science and Technology, Government of India (Unknown); Jawaharlal Nehru Medical College (Other)
Responsible Party: Principal Investigator, Dr. Shweta Khandelwal, Senior Public Health Nutritionist, Centre for Chronic Disease Control, India
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SERC/LS-451/2011
Record Dates: First submitted 2012-04-18; First posted 2012-04-19 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Pregnancy
Keywords: DHA; Omega 3 fatty acid; Decosa hexaenoic acid; Pregnancy; Newborn outcome; Supplementation; Birth size; gestational age; India; Randomized controlled trial; RCT
MeSH Terms: interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Docosa-hexaenoic Acid (DHA) (Active Comparator)
  Interventions: Dietary Supplement: Docosa-hexaenoic acid (DHA)
- Placebo (Placebo Comparator): Corn-Soy Oil
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Docosa-hexaenoic acid (DHA) — 400 mg/day of Docosa-hexaenoic Acid (algal DHA) will given to the pregnant women (in the active group) from ≤20 weeks of gestation through delivery.
  Other Names: DHA; Omega 3 fatty acid
  Arms: Docosa-hexaenoic Acid (DHA)
Dietary Supplement: Placebo — 400 mg/day of placebo (corn/soy oil) will be given to the pregnant women from ≤20 weeks of gestation through delivery.
  Other Names: Corn/Soy oil
  Arms: Placebo

SUMMARY:
The 'DHANI randomized controlled trial" seeks to examine the effects of prenatal DHA supplementation on newborn anthropometry where in healthy pregnant will be assigned to receive either 400 mg of DHA or a placebo daily from ≤20 weeks gestation through delivery.

DETAILED DESCRIPTION:
A double-blinded, randomized, placebo controlled trial would be conducted among pregnant women in India to test the effectiveness of supplementing pregnant Indian women with 400 mg/d algal DHA compared to placebo from mid-pregnancy through delivery. Eligible participants would be randomized to receive either 400 mg of DHA or a placebo baseline measures would be taken before the enrollment of the participant in the study. This study would assess the effect of maternal DHA supplementation on:

1. New born anthropometry (birth weight, length and head circumference)
2. New born APGAR score

ELIGIBILITY:
Inclusion Criteria:

* 18 to 35 year old pregnant women (singleton) at <=20 weeks of gestation (calculated from the LMP by study physician).
* Willing to participate in the study and perform all measurements for self, husband and the offspring including anthropometry, dietary assessment, questionnaires and biological samples (blood and breast milk).
* Willing to provide signed and dated informed consent.

Exclusion Criteria:

* Women allergic (if aware) to any of the test products.
* Women at high risk for hemorrhagic bleeding, clotting (if aware).
* Women with high-risk pregnancies (history and prevalence of pregnancy complications, including abruptio placentae, preeclampsia, pregnancy-induced hypertension, any serious bleeding episode in the current pregnancy, and/ or physician referral); and/or diagnosed chronic degenerative disease(s) such as diagnosed heart disease, cancer, stroke or diabetes (as omega-3 could raise blood sugar and lower insulin production).
* Women consuming omega-3 supplements or having used these in 3 months preceding the intervention period.
* Reported participation in another biomedical trial 3 months before the start of the study or during the study (not to get the results of the present study contaminated).

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 600 (Actual)
Dates: Start 2015-12; Primary Completion 2016-12-06 (Actual); Study Completion 2016-12-09 (Actual)

PRIMARY OUTCOMES:
Newborn anthropometry. | At delivery
  Measures for new born anthropometry would include birth weight, length and head circumference

SECONDARY OUTCOMES:
Gestational age | At delivery
New born APGAR Score | At delivery (1 min and 5 mins)
  APGAR : Appearance, Pulse, Grimace, Activity, Respiration scores
Unfavorable pregnancy outcomes | At delivery
  Still births, low birth weight babies and preterm babies

CONTACTS AND LOCATIONS:
Overall Officials: Shweta Khandelwal, PhD, Principal Investigator — Centre for Chronic Disease Control (CCDC)
Locations (1):
- KLEUs Jawaharlal Nehru Medical College- Prabhakar Kore Charitable Hospital, Belagavi, Karnataka, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khandelwal S, Swamy MK, Patil K, Kondal D, Chaudhry M, Gupta R, Divan G, Kamate M, Ramakrishnan L, Bellad MB, Gan A, Kodkany BS, Martorell R, Srinath Reddy K, Prabhakaran D, Ramakrishnan U, Tandon N, Stein AD. The impact of DocosaHexaenoic Acid supplementation during pregnancy and lactation on Neurodevelopment of the offspring in India (DHANI): trial protocol. BMC Pediatr. 2018 Aug 4;18(1):261. doi: 10.1186/s12887-018-1225-5. PMID 30077178